CLINICAL TRIAL: NCT06012747
Title: Pain After Cesarean Section - A Danish Multicenter Cohort Study.
Status: Completed | Type: Observational
Sponsor: Nordsjaellands Hospital (Other)
Responsible Party: Principal Investigator, Patricia Duch, MD Patricia Duch, Nordsjaellands Hospital
Other Study IDs: 100
Record Dates: First submitted 2023-05-10; First posted 2023-08-25 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Pain; Cesarean Section; Recovery
Keywords: Pain; Cesarean Section; Recovery; REDCap
MeSH Terms: conditions — Pain | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — The patients receive a questionnaire every 6 hours during the first 24 hours after their cesarean section, and again after 2, 7, and 30 days.

SUMMARY:
Pain after a cesarean section is of moderate to severe intensity. A Danish multicenter study from 2021 used an obstetric Quality of Recovery score 24 hours after the cesarean section and found that 45% of 861 patients had experienced very severe pain during recovery.

This result was surprisingly high but also unspecific. Therefore, the investigators aim to investigate the intensity of pain experienced by patients at specific time intervals after the cesarean section e.g., every 6th hour. Additionally, the investigators will examine whether the pain has an impact on important functions for both the patients and the newborns, as well as assess the overall morphine consumption.

All Danish regions have approved the REDCap database as a secure way to collect and store data. REDCap can also send encrypted links that can be converted into SMS messages sent to the participants' mobile phones at fixed intervals, allowing participants to enter data directly into the secure system. The investigators also aim to feasibility test the system.

When a child is delivered by cesarean section, it is an expectation that the mother can take care of herself and the baby a few hours after the surgery. However, severe pain can hinder this. Therefore, it is important to investigate whether pain relief for our patients is sufficient.

Based on response rates and the frequency of outcomes, data from this observational study can support the design of a future national multicenter randomized controlled trial (RCT) with a focus on postoperative pain intervention. The incidences of binary outcome measures and standard deviations of continuous outcome measures will support the sample size calculations for our RCT.

ELIGIBILITY:
Inclusion Criteria Patients who undergo planned cesarean section under spinal anesthesia. Patients must be able to answer a Danish questionnaire via SMS on their phone and provide consent.

Exclusion Criteria:

Age < 18 years

Ages: 18 Years to 50 Years | Sex: Female
Age Groups: Adult
Study Population: Danish patients > 18 years old who undergo planned cesarean section under spinal anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 752 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Self reported pain on movement from supine position to sitting position after 24 hours, NRS 0-10 | 24 hours after cesarean section
  Patient reported
Composite outcome of self reported morphine side effects occurring within 24 hours For vomiting and urinary retention, this is recorded as yes/no, where yes is considered a side effect. | 24 hours after cesarean section
  consisting of either nausea, dizziness, itching, vomiting, or urinary retention.
  Nausea, itching, and dizziness are recorded on a 4-point scale: None, mild, moderate, severe. Where moderate and severe are considered side effects.
  For vomiting and urinary retention, this is recorded as yes/no, where yes is considered a side effect.
Neonatal admission , | within 24 hours
  yes/no

SECONDARY OUTCOMES:
See protokol for the multible secondary and exploratory outcomes | 0-30 days
  See protokol for the multible secondary and exploratory outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Duch, MD, Principal Investigator — Hillerod Hospital, Denmark; Helene Nedergaard, MD, Ph.D, Study Chair — Kolding Sygehus
Locations (19):
- Denmark (19):
  - Department of Anesthesia, Åbenrå Hospital, Aabenraa
  - Department of Anesthesia, Aalborg University Hospital, Aalborg
  - Department of Anesthesia, Århus University Hospital, Aarhus
  - Department of Anesthesia, Copenhagen University Hospital, Rigshospitalet, Copenhagen
  - Department of Anesthesia, Esbjerg Hospital, Esbjerg
  - Department of Anesthesia, Gødstrup Hospital, Gødstrup
  - Department of Anesthesiology, Copenhagen University Hospital, Herlev, Herlev
  - Department of Anesthesiology, Copenhagen University Hospital, North Zealand Hillerød, Hillerød
  - Department of Anesthesia, Hjørring Sygehus, Hjørring
  - Department of Anesthesia, Holbæk Hospital, Holbæk
  - Department of Anesthesia, Horsens Hospital, Horsens
  - Department of Anesthesiology, Copenhagen university Hospital, Hvidovre, Hvidovre
  - Department of Anesthesia and Intensive care, University Hospital of Southern Denmark, Kolding, Kolding
  - Department of Anesthesia, Nykøbing Falster Hospital, Nykøbing Falster
  - Department of Anesthesia, Odense University Hospital, Odense
  - Department of anesthesia, Randers Sygehus, Randers
  - Department of Anesthesia, Zealand University Hospital, Roskilde, Roskilde
  - Department of Anesthesia, Slagelse Hospital, Slagelse
  - Department of Anesthesia,Viborg, Regional Hospital, Viborg

IPD SHARING:
Plan to Share IPD: Undecided
Each participating site has access to the data, which can be viewed by the project managers. Once all the data is collected, it will be anonymized and used for calculations. After the data is published, each participating site can have control over its own data but can only publish it with the permission of the project managers.

REFERENCES:
- [Derived] Duch P, Wikkelso A, Jorgensen CC, Jakobsen JC, Mathiesen O, Norskov AK, Nedergaard H; on the behalf of the National Pain after Cesarean Section (PACS) Working Group . And in collaboration with CEPRA a consortium initiative for peri-operative research (www.cepra.nu). Pain and adverse effects after caesarean delivery: A nationwide prospective cohort study. Eur J Anaesthesiol. 2026 Jan 1;43(1):34-44. doi: 10.1097/EJA.0000000000002277. Epub 2025 Sep 22. PMID 40956058

DOCUMENTS (1):
  • Study Protocol (2023-08-11): https://cdn.clinicaltrials.gov/large-docs/47/NCT06012747/Prot_000.pdf